CLINICAL TRIAL: NCT01003093
Title: A Safety and Immunogenicity Phase 1 Trial With an Adjuvanted TB Subunit Vaccine (Ag85B-ESAT-6 + IC31) Administered at 0 and 2 Months
Brief Title: A Safety and Immunogenicity Trial With an Adjuvanted Tuberculosis(TB) Subunit Vaccine
Acronym: THYB-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THYB-01; Eudract number: TEST-001599-14
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Ag85B; ESAT-6; IC31
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antigen group + high adjuvans (Experimental): The antigen group + high adjuvans group received two injections of antigen (Ag85B + ESAT-6) + IC31 (500 nmol KLK + 20 nmol ODN1a) two months apart.
  Interventions: Biological: 50 microgram antigen (Ag85B + ESAT-6) + 500 nmol KLK + 20 nmol ODN1a
- Antigen group (Experimental): The antigen group received two injections of antigen (Ag85B + ESAT-6) two months apart.
  Interventions: Biological: 50 microgram antigen (Ag85B + ESAT-6)
- Antigen + low adjuvans group (Experimental): The antigen group + low adjuvans group received two injections of antigen (Ag85B + ESAT-6) + IC31 (100 nmol KLK + 4 nmol ODN1a) two months apart.
  Interventions: Biological: 50 microgram antigen (Ag85B + ESAT-6) + 100 nmol KLK + 4 nmol ODN1a

INTERVENTIONS:
Biological: 50 microgram antigen (Ag85B + ESAT-6) — 0.5 mL suspension for injection x 2 with 2 months interval
  Other Names: Antigen H1
  Arms: Antigen group
Biological: 50 microgram antigen (Ag85B + ESAT-6) + 100 nmol KLK + 4 nmol ODN1a — 0.5 mL suspension for injection x 2 with 2 months interval
  Other Names: Antigen H1 + IC31
  Arms: Antigen + low adjuvans group
Biological: 50 microgram antigen (Ag85B + ESAT-6) + 500 nmol KLK + 20 nmol ODN1a — 0.5 mL suspension for injection x 2 with 2 months interval
  Other Names: Antigen H1 + IC31
  Arms: Antigen group + high adjuvans

SUMMARY:
The purpose of this study is to evaluate the safety profile of an adjuvanted TB subunit vaccine administered at 0 and 2 months in healthy BCG-unvaccinated volunteers with no prior history of TB disease or known prior exposure to TB

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy based on medical examination/history at the inclusion
* Age between 18 and 55 years
* Signed informed consent
* Prepared to grant authorized persons access to the medical records
* The volunteer is likely to comply with instructions

Exclusion Criteria:

* Known exposure to TB before (or expected during) the trial
* Prior BCG vaccination
* Granulomatous disease (by chest X-ray, autoimmune screen)
* Vaccinated with live vaccine 3 months before first vaccination
* Administration of immune modulating drugs (steroids, immunosuppressive drugs or immunoglobulins) 3 months before the first vaccination
* HBV, HCV or HIV sero-positive (HBsAg, HBsAb, HBc total and IgM ab and HCV, HIV-1 and HIV2 ab)
* Participation in other clinical trials
* Positive Mantoux or QuantiFERON-TB Gold
* Known hypersensitivity to any of the vaccine components
* Laboratory parameters outside of normal ranges considered clinically relevant

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Physical examination. Local adverse events. Systemic adverse events. Laboratory safety tests including urine safety tests. | From the first vaccination until 8 months after the first vaccination

SECONDARY OUTCOMES:
Detection by ELISPOT of IFN gamma spot-forming cells in PBMC. Detection by ELISA of IFN gamma production in supernatants of PBMC. Detection of humoral response (IgG) by ELISA. | From first vaccination until 36 months after first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jaap van Dissel, MD, Prof., Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, RC Leiden, Netherlands

REFERENCES:
- [Derived] Ottenhoff TH, Doherty TM, van Dissel JT, Bang P, Lingnau K, Kromann I, Andersen P. First in humans: a new molecularly defined vaccine shows excellent safety and strong induction of long-lived Mycobacterium tuberculosis-specific Th1-cell like responses. Hum Vaccin. 2010 Dec;6(12):1007-15. doi: 10.4161/hv.6.12.13143. Epub 2010 Dec 1. PMID 21178394
- [Derived] van Dissel JT, Arend SM, Prins C, Bang P, Tingskov PN, Lingnau K, Nouta J, Klein MR, Rosenkrands I, Ottenhoff TH, Kromann I, Doherty TM, Andersen P. Ag85B-ESAT-6 adjuvanted with IC31 promotes strong and long-lived Mycobacterium tuberculosis specific T cell responses in naive human volunteers. Vaccine. 2010 Apr 30;28(20):3571-81. doi: 10.1016/j.vaccine.2010.02.094. Epub 2010 Mar 11. PMID 20226890